CLINICAL TRIAL: NCT03051243
Title: Safety and Efficacy of Linagliptin Therapy in the Setting of Internal Medicine Department Type 2 Diabetes Mellitus
Brief Title: Safety and Efficiency of Linagliptin (Trajenta) in the Setting of Internal Medicine Department
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Dror Dicker, Head of internal medicine D' and obesity clinic, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0643-14RMC
Record Dates: First submitted 2017-01-15; First posted 2017-02-13 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: DM2
MeSH Terms: interventions — Linagliptin; Insulin Glargine; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linagliptin and Basal Insulin (Active Comparator): linagliptin (trajenta) 5mg once daily combined with basal insulin (glargine Lantus; sanofi) 0.15-0.3 units/kg TDD before bed time.
  Interventions: Drug: Linagliptin and Basal Insulin
- Basal Insulin and Bolus Insulin (Active Comparator): Basal Insulin (Glargine Lantus; Sanofi) based therapy once daily before bedtime and glulisine (Apidra; sanofi) before meals. insulin dose will be 0.5 units/kg divided half as insulin glargine once daily and half as insulin glulisine before meals.
  Interventions: Drug: Basal Insulin and Bolus Insulin

INTERVENTIONS:
Drug: Linagliptin and Basal Insulin — Linagliptin and bed time insulin glargine linagliptin (trajenta) once daily combined with bed time basal insulin (glargine Lantus; sanofi) before meals
  Other Names: Trajenta (Linagliptin)
  Arms: Linagliptin and Basal Insulin
Drug: Basal Insulin and Bolus Insulin — Basal bolus insulin regimen and insulin based therapy with glargine once daily before bedtime and glulisine (Apidra; sanofi) before meals
  Other Names: glargine; glulisine
  Arms: Basal Insulin and Bolus Insulin

SUMMARY:
Prospective, open labels, randomized study. A total of 60 admitted patient between 18 and 85 years old with known with history of DM for more than 3 months and an average of two consecutive blood glucose levels above 180 mg/dl (after stopping all previous oral antidiabetic and insulin on admission) will be enrolled Patient will be randomized to a 1:1 ratio in two treatment groups regimens- linagliptin (trajenta) once daily combined with basal insulin at bed time (glargine Lantus; sanofi) and basal bolus insulin with glargine once daily and glulisine (Apidra; sanifi) before meals.

Patient will be discharged according to discharged protocol. Follow-up visits will take place at 3 and 6 months post discharged.

DETAILED DESCRIPTION:
patient in the linagliptin plus basal insulin will receive linagliptin at single dose of 5 mg/day, and a starting total daily dose (TDD) of glargine of 0.3 units/kg/day, while patients >70 years of age and/or with a serum creatinine >2.0 mg/dL will receive starting TDD of 0.15 units/kg.

Patient in the basal bolus group will start at a TDD of 0.5 units/kg divided half as insulin glargine once daily and half as insulin glulisine before meals. In patients >70 years of age and/or with a serum creatinine >2.0 mg/dL, the starting TDD will be reduce to 0.3 units/kg.

The results of BG values will be measured as 2 hour pre meal glucose, bedtime glucose, and mean daily BG after first day at hospital, HbA1c will be measured on the first day of hospitalization.

Patient with pre-meal and bed time blood glucose levels over 180 mg/dl will receive correctional doses of short acting insulin based on glucose levels as follow- 180-250mg/dl 2 units of insulin, 250-300 mg/dl 3 units of insulin, 350-400 4 units of insulin.

Hypoglycemic events shall be documented as well. In case of treatment failure, defined as average blood glucose levels or two consecutive measurements of more than 240 mg/dl, patient's treatment will be changed to basal based regimen.Patient with pre-meal and bed time blood glucose levels over 180 mg/dl will receive correctional doses of short acting insulin based on glucose levels as follow- 180-250mg/dl 2 units of insulin, 250-300 mg/dl 3 units of insulin, 350-400 4 units of insulin.

Hypoglycemic events shall be documented as well. In case of treatment failure, defined as average blood glucose levels or two consecutive measurements of more than 240 mg/dl, patient's treatment will be changed to basal based regimen.

Patient will be discharged according to discharged protocol. Follow-up visits will take place at 3 and 6 months post discharged.

Patients will be instructed to measure and record BG levels (pre meal glucose, bedtime glucose, and mean daily BG) during three days before follow-ups visits.

ELIGIBILITY:
Inclusion Criteria:

* Male & female patient with Known history of DM for more than 3 months before randomization.
* Hospital admission due to blood glucose levels ranging between 180-400 mg/dl.
* Average of two consecutive blood glucose levels above 180 mg/dl.
* Age between 18 and 85 years old.
* Home treatment with diet alone, any combination of oral antidiabetic agents, or insulin therapy at daily dose <0.4 units/kg.

Exclusion Criteria:

* BG >400 mg/dl in the period before randomization.
* Prior history of hyperglycemic crises.
* Have hyperglycemia without history of diabetes.
* Patient who expected ICU admission or cardiac surgery.
* A history of pancreatitis, active gallbladder disease, Corticosteroid therapy or hepatic disease.
* Impaired renal function (glomerular filtration rate [GFR] <30 mL/min or serum creatinine ≥3.0 mg/dL).
* History of diabetic ketoacidosis.
* Pregnancy.
* Inability to give informed consent (poor mental status).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-11-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patient with mean blood glucose levels | After firts day from admission and Up to 14 days, 3 and 6 month after discharge.
  between 80-180 mg/dl.

SECONDARY OUTCOMES:
Difference in BG values within range | After firts day from admission and Up to 14 days, 3 and 6 month after discharge
  140-180 mg/dl.
Number of hypoglycemic events (BG <70 and or < 40 mg/dL). | After firts day from admission and Up to 14 days, 3 and 6 month after discharge
  <70 and or < 40 mg/dL
Number of episodes of hyperglycemia | After firts day from admission and Up to 14 days, 3 and 6 month after discharge
  >240 mg/dL
TTD (total daily dose) of insulin | After firts day from admission and Up to 14 days, 3 and 6 month after discharge
  units of insulin

IPD SHARING:
Plan to Share IPD: Undecided